CLINICAL TRIAL: NCT00581932
Title: Relationship Between Neurotransmitter Receptor Polymorphisms, Plasma Concentrations and Clinical Response to Clozapine
Status: Completed | Type: Observational
Sponsor: Delwyn D. Miller (Other)
Responsible Party: Sponsor-Investigator, Delwyn D. Miller, Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 199901018
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Schizophrenia
Keywords: clozapine, schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: One group, all subjects with DSM-IV diagnosis of Schizophrenia, age 18-65 who are initiating clozapine therapy.

SUMMARY:
This is a study designed to identify genetic polymorphisms (also called allelic variants or genetic markers) that are associated with response to clozapine. This information will be used to enhance the understanding of clozapine response and side effects. DNA from patients will be examined for significant associations between allelic variants in candidate genes in relation to clozapine effects on positive and negative symptoms, global response, quality of life, relapse rates and side effects.

DETAILED DESCRIPTION:
Patients age 18-65 with a DSM IV diagnosis of schizophrenia who have a history of nonresponse to conventional atypical antipsychotics and who are to be treated with clozapine by their psychiatrist, will be asked to participate at or near the time clozapine therapy is initiated. The Brief Psychiatric Rating Scale (BPRS), Scale for the Assessment of Negative Symptoms (SANS), and the Scale for the Assessment of Positive Symptoms (SAPS) will be performed on all subjects at entry into the study, at 3 weeks, 5 weeks, 8 weeks, and at 4 and 6 months. Adverse effects will be monitored with the Simpson-Angus Scale, Barnes Akathisia scale and the AIMS at each of these time points. The Calgary Depression Scale will also be administered at each visit. A complete neurocognitive assessment battery will be completed at entry and at 6 months for those subjects willing to undergo neurocognitive testing. It is anticipated not all subjects will complete neurocognitive testing. A blood or cheek swab sample will be collected at study entry for DNA analysis. Plasma blood levels will be collected at weeks 3, 5, 8 and study completion for measurement of clozapine plasma concentrations. The subject's weight, BMI, smoking status and concomitant medications will be recorded at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia
* Beginning clozapine therapy
* age 18-65
* must be willing to participate in interviews and provide a DNA sample

Exclusion Criteria:

* no longer taking clozapine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psychiatric clinic, Inpatient Psychiatry unit
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2001-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Brief Psychiatric Rating Scale | entry, 3 wks, 5 wks, 8 wks, 4 mo, 6 mo

SECONDARY OUTCOMES:
Scale for the Assessment of Positive Symptoms | entry, wk 3, wk 5, wk 8, 4 mo, 6 mo
Scale for the assessment of Negative symptoms | entry, 3 wk, 5 wk, 8 wk, 4 mo, 6 mo
Calgary Depression Scale | entry, 3 wk, 5 wk, 8 wk, 4 mo, 6 mo
Abnormal Involuntary Movement Scale | entry, 3 wk, 5 wk, 8 wk, 4 mo, 6 mo
Barnes Akathisia Scale | entry, 3 wk, 5 wk, 8 wk, 4 mo, 6 mo

CONTACTS AND LOCATIONS:
Overall Officials: Del D Miller, PharmD, M.D., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States